CLINICAL TRIAL: NCT07096297
Title: A Phase II Study of Luspatercept Plus Darbepoetin Alfa in Non-mutated SF3B1 Lower-risk Myelodysplastic Syndromes
Brief Title: Luspatercept + Darbepoetin in MDS
Acronym: DarbeLus
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Maximilian Stahl, Assistant Professor, Yale University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000039532
Record Dates: First submitted 2025-07-20; First posted 2025-07-31 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: MDS (Myelodysplastic Syndrome)
Keywords: SF3B1 wild type; RBC transfusion dependent; lower risk; non-mutated SF3B1
MeSH Terms: conditions — Anemia, Refractory, with Excess of Blasts | interventions — luspatercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Luspatercept + Darbepoetin (Experimental): Each participant will be treated with luspatercept every 21 days (three weeks) in combination with darbepoetin alfa every 21 days (three weeks). Both agents will be administered on day 1 of each 21-day cycle. Based on the individual participant's response to combination therapy of luspatercept and darbepoetin alfa, the doses of luspatercept and/or darbepoetin alfa can be either decreased or increased. The starting dose is luspatercept at 1.0 mg/kg (Dose Level 0) and darbepoetin alfa 300 µg (Dose Level 0).
  Interventions: Drug: Luspatercept; Drug: Darbeopoetin

INTERVENTIONS:
Drug: Luspatercept — Luspatercept will be administered every 3 weeks (21 days) at a starting dose of 1.0 mg/kg (Dose Level 0). Luspatercept will be administered to participants by the study staff at the clinical site and administration will be documented in the participant's source record. Participants must have Hgb, blood pressure and weight assessed (changes of body weight of ≤ ± 5% do not require a dose adjustment) prior to each luspatercept dose administration. Subcutaneous injections will be given in the upper arm, thigh, and/or abdomen. Volume for subcutaneous injection will be per institutional standard/guidelines.
Drug: Darbeopoetin — Darbepoetin alfa will be administered every 3 weeks (21 days), at a starting dose of 300 ug (Dose Level 0). Darbepoetin alfa will be administered to participants by the study staff at the clinical site and administration will be documented in the participant's source record. Darbepoetin alfa will be administered as a subcutaneous injection by the site staff in the upper arm, thigh, and/or abdomen per institutional standard/guidelines.

SUMMARY:
This is a single arm open-label Phase II trial of luspatercept and darbepoetin alfa in non-mutated SF3B1 , lower-risk, RBC transfusion dependent MDS participants with an endogenous erythropoietin (EPO) level < 500 IU/L.

DETAILED DESCRIPTION:
This is a single arm open-label Phase II trial of luspatercept and darbepoetin alfa in non-mutated SF3B1 , lower-risk, RBC transfusion dependent MDS participants with an endogenous erythropoietin (EPO) level < 500 IU/L.

Each participant will be treated with luspatercept in combination with darbepoetin alfa every 21 days (three weeks). Both agents will be administered on day 1 of each 21-day (three weeks) cycle. Based on the individual participant's response to combination therapy of luspatercept and darbepoetin alfa, the doses of luspatercept and/or darbepoetin alfa can be either decreased or increased.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and the willingness to sign a written informed consent document.
2. Participant is 18 years or older at the time of signing informed consent.
3. Participant has lower-risk myelodysplastic syndrome (MDS) defined as very low, low and intermediate risk by International Prognostic Scoring System-Revised (IPSS-R) criteria (3).
4. Bone marrow biopsy within 90 days of screening demonstrated less than 5% blasts in the aspirate and/or core biopsy. If no bone marrow biopsy was done within 90 days of screening it is mandatory to repeat it at screening. Otherwise, bone marrow biopsy is optional at screening to obtain correlative study samples.
5. Absence of SF3B1 mutation and del5q.
6. Endogenous serum erythropoietin alfa (EPO) level < 500 IU/L.
7. Participant is transfusion dependent defined as ≥ 2 packed red blood cell (PRBC) units/8 weeks for a minimum of eight weeks immediately prior to screening. The maximum consecutive timeframe participants may be RBC transfusion-free within this 8-week time period is six weeks.

   a. Red blood cell transfusions administered when hemoglobin levels were > 9.0 g/dL and/or RBC transfusions administered for elective surgery, infections or bleeding events will not be counted in above.
8. Participant has an Eastern Cooperative Oncology Group (ECOG) performance status of 0-3 (Appendix 1. ECOG Performance Status Scale).
9. Participant has adequate organ function defined as:

   1. Serum aspartate aminotransferase/serum glutamic oxaloacetic transaminase (AST/SGOT) and alanine aminotransferase (ALT/SGPT) ≤ 3 x ULN, unless considered due to organ involvement by the participant's myeloid malignancy (in that case a cut off ≤ 5 x ULN will be used).
   2. Serum direct bilirubin < 1.5 x ULN.
   3. Creatinine clearance > 30 mL/min based on the Cockroft-Gault glomerular filtration rate (GFR) estimation.
10. Participants must adhere to the following reproductive and contraceptive requirements while on study treatment and for three months after the last dose of luspatercept and darbepoetin alfa:

    a. General Requirements: i. Participants must not be pregnant or breastfeeding. ii. Participants must not donate gametes (i.e., eggs or sperm) or freeze gametes for future use related to assisted reproduction.

    b. For participants of childbearing potential: i. Participant of childbearing potential is defined as an individual who is premenopausal and capable of becoming pregnant, including those using contraception, those who are single, or those with partners who have had a vasectomy.

ii. A negative highly sensitive pregnancy test must be obtained at screening, and a negative serum or urine pregnancy test must be obtained within 72 hours starting on treatment, and participants must agree to further pregnancy tests throughout the study as required per the site's institutional guidelines.

iii. Participants must agree to use two methods of contraception of which one must be highly effective for three months after the last dose of luspatercept and darbepoetin alfa.

c. For Partners of Participants: i. If the participant's partner is of childbearing potential, the partner must also practice a highly effective method of contraception while the participant is on study treatment and for three months after the last dose of luspatercept and darbepoetin alfa, unless the participant is vasectomized.

d. Highly effective methods of contraception include, but are not limited to: i. Combined hormonal contraception (estrogen and progestogen) that inhibits ovulation (oral, intravaginal, or transdermal).

ii. Progestogen-only hormonal contraception that inhibits ovulation (oral, injectable, or implantable).

iii. Non-hormonal (cooper) intrauterine device (IUD). iv. Intrauterine hormone-releasing system. v. Bilateral tubal occlusion. vi. Sexual abstinence (the reliability of abstinence must be evaluated concerning the duration of the clinical study and the participant's lifestyle).

vii. A vasectomized partner (provided the partner is the sole sexual partner of the study participant of childbearing potential and that the vasectomized partner has received medical confirmation of the surgical success).

Exclusion Criteria:

1. Prior treatment with ESA, luspatercept, hypomethylating agents or lenalidomide/thalidomide/other immunomodulating drug (IMiDs).

   1. Exception 1: Participants can have received ≤ 2 doses of prior epoetin alfa or ≤ 1 dose darbepoetin alfa if ≥ 8 weeks from date of consent.
   2. Exception 2: Participants can have received ≤ 1 week of treatment with lenalidomide ≥ 8 weeks from the date of consent, at the sponsor-investigator's discretion.
   3. After signing consent, the participants are not allowed to receive any of these drugs: other RBC hematopoietic growth factors (e.g., Interleukin-3), granulocyte colony stimulating factors (i.e., G-CSF, GM-CSF), except in cases of neutropenic fever, cytotoxic, chemotherapeutic, targeted or investigational agents/therapies, azacitidine, decitabine or other hypomethylating agents, lenalidomide, thalidomide and other immunomodulating drugs (IMiDs), hydroxyurea, androgens, unless to treat hypogonadism, oral retinoids (topical retinoids are permitted), arsenic trioxide, interferon and interleukins.
2. Participants with history of seizures at any time.
3. Participants with any of the following conditions within six months prior to screening:

   1. Stroke.
   2. Thrombosis/thromboembolism.
   3. Myocardial infarction.
   4. Uncontrolled angina.
   5. Acute decompensated cardiac failure or New York Heart Association (NYHA) Class III-IV heart failure.
   6. Uncontrolled cardiac arrhythmia as determined by the investigator.
4. Participant has immediate life-threatening, severe complications of their myeloid malignancy such as uncontrolled bleeding, pneumonia with hypoxia or shock, and/or disseminated intravascular coagulation.
5. Participants with uncontrolled hypertension defined as systolic blood pressure (SBP) of ≥ 150 mmHg and/or diastolic blood pressure (DBP) ≥ 100 mmHg despite adequate treatment. Participant with history of cerebrovascular accident (including ischemic, embolic, and hemorrhagic cerebrovascular accident), transient ischemic attack.
6. Participant has active viral infection with human immunodeficiency virus (HIV), or active infection with hepatitis B virus (HBV) or active infection with hepatitis C virus (HCV). Participants with HIV that is controlled (not detectable viral load) with highly active antiretroviral therapy (HAART) are eligible to participate.
7. Participant has active uncontrolled systemic fungal, bacterial, or viral infection (defined as ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics, antiviral therapy, and/or other treatment).
8. Participant who is pregnant or lactating.

   1. Pregnant participants are excluded from this study because luspatercept has shown in animal studies to be potentially associated with fetal harm.
   2. Because there is an unknown but potential risk for AE in nursing infants secondary to treatment, lactating participants are excluded from this study.
9. Participant with prior history of malignancies, other than MDS, unless the participant has been free of the disease for ≥ 5 years. However, participants with the following history/concurrent conditions are allowed:

   1. Basal or squamous cell carcinoma of the skin.
   2. Carcinoma in situ of the cervix.
   3. Carcinoma in situ of the breast.
   4. Incidental histologic finding of prostate cancer (T1a or T1b using the tumor, nodes, metastasis TNM clinical staging system).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2030-08 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
Mean Rate of Red Blood Cell Transfusion Independence | 24 weeks
  Mean rate of red blood cell transfusion independence (RBC-TI) for at least any consecutive 84 days (≥ 12 consecutive weeks) during weeks 1-24 compared to baseline in non-mutated SF3B1, lower-risk myelodysplastic syndrome patients treated with Luspatercept plus Darbepoetin Alfa
Mean Rate of Hemoglobin Increase | 24 weeks
  Mean rate of hemoglobin ≥ 1.5 g/dL during weeks 1-24 compared to baseline in non-mutated SF3B1, lower-risk myelodysplastic syndrome patients treated with Luspatercept plus Darbepoetin Alfa.

SECONDARY OUTCOMES:
Mean rate of Red Blood Cell Transfusion Independence for ≥8 Consecutive Weeks During Weeks 1-24 | 24 weeks
  Mean rate of red blood cell transfusion independence (RBC-TI) for at least 8 consecutive weeks during weeks 1-24 compared to baseline. Assessed as the proportion of participants who achieve RBC-TI within the first 24 weeks of the study.
Mean rate of Red Blood Cell Transfusion Independence for ≥8 Consecutive Weeks During Weeks 1-48 | 48 weeks
  Mean rate of red blood cell transfusion independence (RBC-TI) for at least 8 consecutive weeks during weeks 1-48 compared to baseline. Assessed as the proportion of participants who achieve RBC-TI within the first 48 weeks of the study.
Mean rate of Red Blood Cell Transfusion Independence for ≥12 Consecutive Weeks During Weeks 1-24 | 24 weeks
  Mean rate of red blood cell transfusion independence (RBC-TI) for at least 12 consecutive weeks during weeks 1-24 compared to baseline. Assessed as the proportion of participants who achieve RBC-TI within the first 24 weeks of the study.
Mean rate of Red Blood Cell Transfusion Independence for ≥12 Consecutive Weeks During Weeks 1-48 | 48 weeks
  Mean rate of red blood cell transfusion independence (RBC-TI) for at least 12 consecutive weeks during weeks 1-48 compared to baseline. Assessed as the proportion of participants who achieve RBC-TI within the first 48 weeks of the study.
Mean rate of Red Blood Cell Transfusion Independence for ≥24 Consecutive Weeks During Weeks 1-24 | 24 weeks
  Mean rate of red blood cell transfusion independence (RBC-TI) for at least 24 consecutive weeks during weeks 1-24 compared to baseline. Assessed as the proportion of participants who achieve RBC-TI within the first 24 weeks of the study.
Mean rate of Red Blood Cell Transfusion Independence for ≥24 Consecutive Weeks During Weeks 1-48 | 48 weeks
  Mean rate of red blood cell transfusion independence (RBC-TI) for at least 24 consecutive weeks during weeks 1-48 compared to baseline. Assessed as the proportion of participants who achieve RBC-TI within the first 48 weeks of the study.
Duration of Red Blood Cell Transfusion Independence for ≥8 Weeks | Assessed throughout the entire study period, approximately 2.5 years
  To determine the duration of red blood cell transfusion independence (RBC-TI) for at least 8 consecutive weeks. This outcome measure will evaluate how long participants maintain RBC-TI for a minimum of 8 weeks during the study period.
Duration of Red Blood Cell Transfusion Independence for ≥12 Weeks | Assessed throughout the entire study period, approximately 2.5 years
  Duration of red blood cell transfusion independence (RBC-TI) for at least 12 consecutive weeks. Assessed as how long participants maintain RBC-TI for a minimum of 12 weeks during the study period.
Duration of Red Blood Cell Transfusion Independence for ≥24 Weeks | Assessed throughout the entire study period, approximately 2.5 years
  To determine the duration of red blood cell transfusion independence (RBC-TI) for at least 24 consecutive weeks. Assessed as how long participants maintain RBC-TI for a minimum of 24 weeks during the study period.
Median Time to Red Blood Cell Transfusion Independence for ≥8 Consecutive Weeks | Assessed throughout the entire study period, approximately 2.5 years
  Median time to achieve red blood cell transfusion independence (RBC-TI) for at least 8 consecutive weeks. Assessed as the median duration of time it takes for participants to achieve RBC-TI for a minimum of 8 weeks during the study period.
Median Time to Red Blood Cell Transfusion Independence for ≥12 Consecutive Weeks | Assessed throughout the entire study period, approximately 2.5 years
  Median time to achieve red blood cell transfusion independence (RBC-TI) for at least 12 consecutive weeks. Assessed as the median duration of time it takes for participants to achieve RBC-TI for a minimum of 12 weeks during the study period.
Median Time to Red Blood Cell Transfusion Independence for ≥24 Consecutive Weeks | Assessed throughout the entire study period, approximately 2.5 years
  Median time to achieve red blood cell transfusion independence (RBC-TI) for at least 24 consecutive weeks. Assessed as the median duration of time it takes for participants to achieve RBC-TI for a minimum of 24 weeks during the study period.
Mean rate of Hematological Improvement Based on MDS 2018 IWG Response Criteria | Assessed throughout the entire study period, approximately 2.5 years
  Mean rate of hematological improvement (HI) in participants as defined by the Myelodysplastic Syndromes (MDS) 2018 International Working Group (IWG) response criteria.
Changes in Health-Related Quality of Life (HRQoL) Using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) | At baseline, every 21 days during the treatment period, during the 24 week response assessment (approximately 169 days after beginning study treatment), at the end of treatment visit and during the 42 day follow up visit
  Health-related quality of life (HRQoL) will be assessed using the EORTC QLQ-C30. This outcome measure will evaluate participants' overall quality of life, functional status, and symptom burden at various time points throughout the study. Scoring Range: 0 to 100 for each scale. Functioning Scales: Higher scores = better functioning. Symptom Scales: Higher scores = worse symptoms. Global Health Status/QOL Scale: Higher scores = better overall QOL.
Changes in Anemia Outcome Measures Using the Functional Assessment of Cancer Therapy - Anemia (FACT-An) Questionnaire | At baseline, every 21 days during the treatment period, during the 24 week response assessment (approximately 169 days after beginning study treatment), at the end of treatment visit and during the 42 day follow up visit
  Changes in anemia-related quality of life using the FACT-An questionnaire. This outcome measure will evaluate the impact of anemia on participants' well-being, including physical, social, and emotional functioning, at various time points throughout the study. Scoring Range: 0 to 188 total. Higher scores=better QOL.
Changes in Quality of Life Using the Quality of Life in Myelodysplasia Scale (QUALMS-P) Questionnaire | At baseline, every 21 days during the treatment period, during the 24 week response assessment (approximately 169 days after beginning study treatment), at the end of treatment visit and during the 42 day follow up visit
  Changes in quality of life specific to myelodysplasia using the QUALMS-P questionnaire. This outcome measure will evaluate the effects of myelodysplasia on participants' day-to-day life and overall well-being at various time points throughout the study. Total score 0-100. Higher scores=better QOL.

CONTACTS AND LOCATIONS:
Overall Officials: Maximilian Stahl, MD, Principal Investigator — Yale University
Locations (3):
- United States (3):
  - Yale University, New Haven, Connecticut
  - Robert H. Lurie Comprehensive Cancer Center of Northwestern University, Chicago, Illinois
  - Harold C. Simmons Comprehensive Cancer Center of UT Southwestern, Dallas, Texas